CLINICAL TRIAL: NCT01529476
Title: A Randomized, Double-Blind, Comparative, Multi-Center Study of the Safety and Efficacy of TG-873870(Nemonoxacin) Versus Levofloxacin in Adult Patients With Community-Acquired Pneumonia (CAP)
Brief Title: Study to Evaluate the Efficacy and Safety of Oral Administration With Nemonoxacin and Levofloxacin in Patients With CAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Collaborators: Qualitix Clinical Research Co., Ltd. (Industry); Parexel (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-873870-C-4
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Pneumonia
Keywords: Ofloxacin; Levofloxacin; Ofloxacin hydrochloride
MeSH Terms: conditions — Pneumonia | interventions — Levofloxacin; nemonoxacin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nemonoxacin 500 mg (Experimental)
  Interventions: Drug: Nemonoxacin
- Levofloxacin 500 mg (Active Comparator)
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin — levofloxacin 500 mg,QD,7~10 days
  Arms: Levofloxacin 500 mg
Drug: Nemonoxacin — Nemonoxacin 500mg,QD,7~10 days
  Arms: Nemonoxacin 500 mg

SUMMARY:
1. This study will test the safety and efficacy of TG-873870 (Nemonoxacin) compared with Levofloxacin in adult patients with Community-Aquired Pneumonia (CAP)
2. To investigate the population pharmacokinetics (PPK) of nemonoxacin in adult patients with CAP after continuous oral administration and determine the pharmacokinetic (PK)/pharmacodynamic (PD).

DETAILED DESCRIPTION:
Community-acquired Pneumonia (CAP) remains a leading cause of death in both developing and developed countries. In the choice of antibacterial agents used to treat CAP, fluoroquinolones have received considerable attention because of their wide spectrum of bactericidal activity. TG-873870 (Nemonoxacin), a non-fluorinated quinolone (NFQ), is a selective bacterial topoisomerase inhibitor. This study will test the safety and efficacy of TG-873870 (Nemonoxacin) compared with Levofloxacin in adult patients with Community-Aquired Pneumonia (CAP).

Besides,the population pharmacokinetics (PPK) of nemonoxacin in adult patients with CAP after continuous oral administration and determine the pharmacokinetic (PK)/pharmacodynamic (PD).

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 70;
2. Weighs between 40 ~ 100 kg, and BMI ≥ 18 kg/m2;
3. Must have a clinical diagnosis of CAP
4. Chest X-ray shows new or persist/progressive infiltrates
5. If female, non-lactating and at no risk or pregnancy (post-menopausal or must use adequate birth control)
6. The patient is able to take the drug orally.

Exclusion Criteria:

1. Patients with CAP that, in the investigator's judgment, is severe enough to require hospitalization for intravenous antibiotic therapy and/or supplemental oxygen therapy with ICU support
2. Known or suspected severe bronchiectasis, cystic fibrosis, active pulmonary tuberculosis or infection with other mycobacteria or fungi, known bronchial obstruction, a history of post-obstructive pneumonia, other confounding respiratory diseases, such as lung cancer, malignancy metastatic to the lungs, lung abscess, empyema, suspected aspiration pneumonia due to vomiting, or non-bacterial respiratory infection (chronic obstructive pulmonary disease [COPD] is not exclusionary)
3. Clinically significant conduction or other abnormality on 12-lead ECG, or QTc interval
4. Potassium is < 3.5 mmol/L
5. Any known disease that seriously affect the immune system
6. Active hepatitis or decompensated cirrhosis;
7. Have used quinolones or fluoroquinolones within 14 days before enrollment
8. Patients who are being or will be on a long-term medication of steroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Per subject clinical cure rate | 21days
  The clinical cure rate will be evaluated according to signs and symptoms and changes in the chest X-ray.

SECONDARY OUTCOMES:
Safety Evaluation | 24days
  Clinical adverse events and abnormal laboratory or other special test findings during this study should be observed and recorded carefully.
Per subject microbiological cure rate | 14 days
  The microbiological cure rate will be evaluated according to the microbiological identification results of the central laboratory
Per subject overall cure rate | 14 days
  Evaluate the overall efficacy after a comprehensive consideration of the clinical results and the bacteriological results.

CONTACTS AND LOCATIONS:
Locations (57):
- China (42):
  - Anzhen Hospital,Beijing Capital Medical University, Anzhen
  - Beijing Union Medical College Hospital, Beijing
  - General Hospital of PLA Second Artillery, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Chaoyang Hospital, Chaoyang
  - West China Hospital of Sichuan University,Center for Infection Disease, Chengdu
  - PLA Third Militrary Medical University,Second Affiliated Hospital, Chongqing
  - PLA Third Militrary Medical University,Third Affiliated Hospital, Chongqing
  - The First Affiliated Hospital,Chongqing Medical University, Chongqing
  - The First Hospital of Fujian Medical University, Fuzhou
  - People's Hospital of Gansu Province, Gansu
  - GuangZhou Red Cross Hospital, Guangzhou
  - Sun Yet-sen Memorial Hospital, Guangzhou
  - Affilated Hospital of Guilin Medical college, Guilin
  - Hainan Provincial People's Hospital, Hainan
  - Hospital Affiliated to Hainan Medical College, Hainan
  - Hubei General Hospital, Hubei
  - Taihe Hospital, Hubei
  - Hunan Provincial People's Hospital, Hunan
  - Third Xiangya Hospital,Central South University, Hunan
  - People's Hospital of Jiangxi Province, Jiangxi
  - Jinan Central Hospital, Jinan
  - Lanzhou university second hospital, Lanzhou
  - Shengjing Hospital of China Medical University, Liaoning
  - Second Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Genrak Hospital of Nanjing Millitary Command, Nanjing
  - Huadong Hospital of Fudan University, Shanghai
  - Putuo Central Hospital, Shanghai
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai East Hospital in Pudong New Area, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - The First Hospital of Shanxi Medical College, Shanxi
  - PLA General Hospital of Shenyang Military Region, Shenyang
  - ShenZhen People's Hospital, Shenzhen
  - Institute of Antibiotics,Huashan Hospital ,Fudan University, Shianghai
  - Department of Resoiratory Medicine,West China Hospital of Sichuan University, Sichuan
  - Shuang Ho Hospital, Taipei
  - The Second Hospital of Wenzhou Medical College, Wenzhou
  - Wuhan General Hospital of Guangzhou Millitary Command, Wuhan
  - The First Affiliated Hospital,Xinjiang Medical University, Xinjiang
  - First Affiliated Hospital,Zhejiang University School of Medicine, Zhejiang
- Taiwan (15):
  - Chia-Yi Christian Hospital, Chiayi City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung hang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Yuan's General Hospital, Kaohsiung City
  - ChiMei Medical Hospital-Liuying branch, Liuying
  - Cheng Ching General Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Veterans General Hospital-TaiChung, Taichung
  - Cheng Hsin General Hospital, Taipei
  - Far-East Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Veterans General Hospital-Taipei, Taipei

REFERENCES:
- [Derived] Yuan J, Mo B, Ma Z, Lv Y, Cheng SL, Yang Y, Tong Z, Wu R, Sun S, Cao Z, Wu J, Zhu D, Chang L, Zhang Y; Investigator Group of the Phase 3 Study on Oral Nemonoxacin. Safety and efficacy of oral nemonoxacin versus levofloxacin in treatment of community-acquired pneumonia: A phase 3, multicenter, randomized, double-blind, double-dummy, active-controlled, non-inferiority trial. J Microbiol Immunol Infect. 2019 Feb;52(1):35-44. doi: 10.1016/j.jmii.2017.07.011. Epub 2017 Aug 2. PMID 30181096